CLINICAL TRIAL: NCT03443674
Title: A Phase I Study Evaluating Safety, Tolerability, and Pharmacokinetics of SCB-313, a Fully-Human TRAIL-Trimer Fusion Protein, for the Treatment of Peritoneal Malignancies
Brief Title: Study With SCB-313 (Recombinant Human TRAIL-Trimer Fusion Protein) for Treatment of Peritoneal Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLO-SCB-313-001
Record Dates: First submitted 2018-01-07; First posted 2018-02-23 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Peritoneal Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCB-313 (Experimental): Dose escalation cohorts--10mg, 20mg, 40mg, 80mg, 160mg. For each cohort: administered twice weekly (eg.. Monday and Thursday or Tuesday and Friday) for 2 weeks (Days 1, 4, 8, and 11) by IP bolus injection.
  Interventions: Drug: SCB-313

INTERVENTIONS:
Drug: SCB-313 — Lyophilized powder in a single-use vial
  Other Names: recombinant human TRAIL-Trimer fusion protein

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, immunogenicity, and PK/PD of SCB-313 (recombinant human TRAIL-Trimer fusion protein) administered twice weekly for 2 weeks via IP bolus injection for the treatment of patients with peritoneal malignancies, including but not limited to peritoneal carcinomatosis, malignant ascites, pseudomyxoma peritonei, and peritoneal mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed peritoneal malignancies after failure or refusal of all approved therapies, and no better option available in the Investigator's opinion.
2. Eastern Cooperative Oncology Group (ECOG) performance status: 0 to 2 (Patients with ECOG score of 3 might be allowed to enter this trial per Investigator's judgment)
3. Life expectancy of at least 8 weeks
4. Age ≥18 years
5. Body mass index ≥17.0 kg/m2
6. Adequate hematological function, defined as:

   1. Platelet count ≥ 75,000/μL
   2. Prothrombin time and activated partial thromboplastin time ≤1.5 times the upper limit of normal (ULN)
   3. Absolute neutrophil count ≥1,500/μL
   4. Hemoglobin ≥8 g/dL (transfusion and erythropoietic agents are allowed. In case there is existence of active bleeding or other persistent condition of either increased destruction or impaired production of erythrocytes which may require repeated transfusion or erythropoietic treatment, the eligibility must be discussed with the Sponsor on a case-by-case basis prior to randomization)
7. Adequate renal function, defined as serum creatinine ≤2.0 times ULN and creatinine clearance >45 mL/minute
8. Adequate liver function, defined as:

   1. Aspartate aminotransferase and alanine aminotransferase ≤3 times ULN for patients without liver metastases, or ≤5 times ULN in the presence of liver metastases
   2. Bilirubin ≤1.5 times ULN, unless patient has known Gilbert's syndrome
9. Female patients of childbearing potential (excluding women who have undergone surgical sterilization or menopause. Menopause is defined as the status where no menstrual periods continue for 1 year or more without any other medical reasons), are eligible if they have negative serum pregnancy testing within 7 days prior to first dosing and are willing to use an effective method of birth control/contraception to prevent pregnancy until 6 months after discontinuation of the SCB-313.

Both men and women of reproductive potential must agree to use effective contraception during the study and for 6 months after discontinuation of the SCB-313.

Note: Contraceptive methods that are considered highly effective are, for example, total abstinence, an intrauterine device, a double barrier method (such as condom plus diaphragm with spermicide), a contraceptive implant, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices, or injections with prolonged release), or have a vasectomized partner with confirmed azoospermia.

Exclusion Criteria:

1. Acute or chronic infection (such as tuberculosis) requiring antiviral or intravenous (IV) antibiotics within 2 weeks prior to enrollment.
2. Symptoms or signs (including laboratory tests) of clinically significant concomitant hematologic, cardiovascular, pulmonary, hepatic, renal, pancreatic, or endocrine diseases.
3. Residual adverse events (AEs) > Grade 2 from previous treatment.
4. Evidence or suspicion of relevant psychiatric impairment including alcohol or recreational drug abuse.
5. Myocardial infarction within 6 months prior to treatment, and/or prior diagnoses of congestive heart failure (New York Heart Association Class III or IV), unstable angina, unstable cardiac arrhythmia requiring medication, and/or long QT syndrome or QT/QTc interval >450 msec at baseline.
6. Uncontrolled hypertension defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg confirmed upon repeated measures.
7. Left ventricular ejection fraction <40% as determined by echocardiography performed at screening or within 90 days prior to enrollment.
8. Prior anti-tumor therapy (chemotherapy) within 2 weeks, hormone therapy or palliative extra-abdominal radiotherapy within at least 1 week, or small-molecule targeted therapy within 5 half-lives prior to enrollment. Prior therapy with monoclonal antibody should be stopped after Investigator's judgement making sure delayed side effects will not interfere with the dose limiting toxicity (DLT) evaluation period after SCB-313 therapy.
9. Major surgery within 4 weeks prior to enrollment.
10. Patient with ileus within 30 days prior to screening.
11. Positive serology test for human immunodeficiency virus Type 1 and 2 or known history of other immunodeficiency disease.
12. Live vaccine within 2 weeks prior to enrollment.
13. Scheduled participation in another clinical study involving an investigational product or device during the course of this study.
14. Previous treatment with a TRAIL-based therapy or death receptor (DR) 4/5 agonist therapy.
15. Known or suspected hypersensitivity to any component of the SCB-313.
16. Any further condition which, according to the Investigator, may result in undue risk of the patient by participating in the present study.
17. Untreated central nervous system metastatic disease, leptomeningeal disease, or cord compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Occurrence of serious adverse events (SAEs) and/or TEAEs | Up to 41 days after start of treatment
  Regardless of causality or relationship to SCB-313 graded using National Cancer Institute Common Terminology Criteria for Adverse Events Version.4.03 (NCI CTCAE v4.03).

SECONDARY OUTCOMES:
Immunogenicity: Occurrence of binding and neutralizing anti-SCB-313 antibodies | Up to 41 days after start of treatment
  Occurrence of binding and neutralizing anti-SCB-313 antibodies
Pharmacokinetics (Cmax) | Up to 12 days after start of treatment
  Maximum serum concentration
Pharmacokinetics (Cmax/D) | Up to 12 days after start of treatment
  Dose-normalized Cmax of SCB-313
Pharmacokinetics (tmax) | Up to 12 days after start of treatment
  Time to Cmax of SCB-313
Pharmacokinetics ([AUC]0-24) | Up to 12 days after start of treatment
  Area under SCB-313 concentration time curve from zero to 24 hours
Pharmacokinetics (AUC0-24/D) | Up to 12 days after start of treatment
  Dose-normalized AUC0-24 of SCB-313
Pharmacokinetics ((AUC0-last)) | Up to 12 days after start of treatment
  Area under curve from time 0 on Day 1 to the last quantifiable concentration time point
Pharmacokinetics (Ctrough) | Up to 12 days after start of treatment
  Trough concentration of SCB-313 at each predose and at 24 hours after the last dose

OTHER OUTCOMES:
CEA | Up to 6 months after start of treatment
  Changes in serum tumor marker（CEA）
Caspase-cleaved cytokeratin 18 (CK-18) | Up to 21 days after start of treatment
  Changes in serum PD biomarkers

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Liverpool Hospital, Liverpool, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - John Flynn Private Hospital, Tugun, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia